CLINICAL TRIAL: NCT04938596
Title: Strengthening of Airborne Preventive Measures Inside Households of Pulmonary TB Cases as a Tool to Reduce New Infections in Close Contacts. A Pilot, Controlled, Pre-post Study.
Brief Title: Airborne Preventive Measures to Reduce New TB Infections in Household Contacts
Acronym: TBMask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government); Agencia Nacional de Investigación y Desarrollo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1211225
Record Dates: First submitted 2021-05-12; First posted 2021-06-24 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Tuberculosis, Pulmonary; Household Contacts; Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis

STUDY DESIGN:
Intervention Model Description: Prospective, semi-experimental, controlled trial.
  Two different health care areas of Santiago (and their corresponding TB clinics) will be allocated to control or intervention arm; after a baseline pre-intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory Bundle Group (Experimental): The intervention consists of a bundle of measures for respiratory transmission prevention that will be provided during the first 2 weeks of TB treatment of index case.
  Interventions: Combination Product: Respiratory bundle
- Standard of care (No Intervention): Under current national guidelines, no systematic recommendation regarding respiratory protection is given for household contacts of TB cases.

INTERVENTIONS:
Combination Product: Respiratory bundle — * Provision of N95 masks and strong recommendation of use to all household contacts and the index case when sharing a room together, for 2 weeks
  * Recommendation to index case to sleep in a room alone, with the door closed and avoid sharing room with others during 2 weeks
  * Promotion of strategies to improve house ventilation during 2 weeks
  * Provision of a TB leaflet and nurse education about TB transmission.
  Arms: Respiratory Bundle Group

SUMMARY:
Tuberculosis (TB) is currently one of the top 10 causes of death worldwide and the leading cause of death from a single infectious agent (ranking above HIV/AIDS). The investigators hypothesize that reducing respiratory exposure within the household, during the first weeks of TB treatment initiation of the index case, can reduce new TB infections in close contacts. For this purpose, a pilot, controlled, pre-post study will be set up, to evaluate the feasibility of implementing a bundle of respiratory precautions to all household contacts of new pulmonary TB cases, compared to standard of care, in primary health care in a high TB incidence area in Santiago, Chile.

DETAILED DESCRIPTION:
Tuberculosis (TB) is currently one of the top 10 causes of death worldwide and the leading cause of death from a single infectious agent (ranking above HIV/AIDS). In 2018, an estimated 10 million people fell ill with TB worldwide, and more than 1.4 million people died from it, making eradication of this disease in the next decades highly unlikely unless new interventions are discovered. Mycobacterium tuberculosis (Mtb) transmission mainly occurs when patients affected by laryngeal or pulmonary TB cough upon others and the mycobacteria are spread in airborne droplets nuclei smaller than 5 μm that are subsequently inhaled by close contacts. Although chemoprophylaxis once a new TB infection is detected is an effective strategy to reduce the risk of contacts developing active TB, it does not prevent Mtb acquisition; it only reduces the risk of developing active TB once infected. Currently, the large majority of international guidelines recommend strict measures to reduce airborne transmission in hospitalized patients with pulmonary TB, with a minimum of 2 weeks of effective TB therapy to consider a patient no longer infectious and discontinue respiratory isolation in healthcare settings. On the contrary, in the community, no special recommendations regarding protection of household contacts are specified, assuming that most of them are already infected and that the TB index case will stop infecting very quickly under antimicrobial treatment. However, several studies show that median time to sputum Mtb culture conversion under effective treatment takes 5-7 weeks, raising the potential for continued transmission even despite effective treatment. Furthermore, a previous study has shown that in Santiago, Chile, 55% of household contacts of TB cases have no evidence of TB infection at the time of diagnosis of the index case - as categorized by negative latent TB testing - yet under close follow-up, up to 21% of these show new evidence of having acquired the infection based on latent TB test conversion after 12 weeks of follow-up. The investigators hypothesize that reducing respiratory exposure within the household, during the first weeks of TB treatment initiation of the index case, can reduce new TB infections in close contacts. For this purpose, a pilot, controlled, pre-post study will be done to evaluate the feasibility of implementing a bundle of respiratory precautions to all household contacts of new pulmonary TB cases, compared to standard of care, in primary care in a high TB incidence area in Santiago. The respiratory bundle in the intervention arm will be implemented as soon as a new pulmonary TB case is diagnosed, will last 2 weeks and, will include: (a) provision of N95 masks and strong recommendation of use to all household contacts and the index case when sharing a room together, (b) recommendation to index case to sleep in a room alone, with the door closed and avoid sharing room with others, (c) promotion of strategies to improve house ventilation; and (d) education about TB transmission. The investigators expect to show that this trial is feasible to proceed with a larger, definitive cluster randomized controlled trial that will evaluate the intervention effectiveness in reducing the incidence of new TB infections in household contacts. The results of this study will help to answer a critical research gap in TB infection control and prevention and, it will provide a key contribution to future policies regarding TB control and elimination worldwide. Furthermore, in the new global context of rising infectious agents of pandemic risk, this work may have an additional potential relevance with respect to the use, acceptability and transmission prevention potential of a respiratory bundle in the household setting regarding other respiratory pathogens such as SARS-Cov-2.

ELIGIBILITY:
Inclusion Criteria:

* all household contacts of a new case of pulmonary TB (smear, culture or PCR positive) newly diagnosed at each clinic.

Exclusion Criteria:

* household contacts found to have co-prevalent active TB at enrolment
* household contacts planning to leave the house at the time of enrolment
* household contacts of index cases having already initiated TB treatment for > 48h
* household contacts of index cases that are currently hospitalized

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Participation rate | 2 weeks
  To document the proportion of TB cases and household contacts who agree to participate as measured by enrollment.
Study compliance | 2 weeks
  To document participants compliance with the respiratory bundle as measured by a previously validated adherence questionnaire.
Completion rate | 12 weeks
  The number of participants assessable at end of follow-up.
Acceptability of the intervention | 12 weeks
  Focus group evaluation (participants and TB nurses perspectives, qualitative outcome).

SECONDARY OUTCOMES:
New tuberculosis infections | 12 weeks
  The number of participants converting from a negative to a positive latent TB test at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: María Elvira Balcells, MD; MSc, Principal Investigator — School of Medicine. Pontificia Universidad Católica de Chile.
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided